CLINICAL TRIAL: NCT00837863
Title: A Twelve Month, Phase II, Randomized, Open-Label, Multi-Center, Dose-Ranging Study of Weekly ALTU-238 (Somatropin) as Compared With Daily Nutropin AQ (Somatropin) in Prepubertal Children With Growth Hormone Deficiency
Brief Title: Study of Weekly ALTU-238 Compared With Daily Nutropin AQ in Prepubertal Children With Growth Hormone Deficiency
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Altus Pharmaceuticals (Industry)
Responsible Party: Kenneth Attie, M.D., Altus Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0001194
Record Dates: First submitted 2009-02-02; First posted 2009-02-05 (Estimated); Last update posted 2009-05-07 (Estimated); Status verified 2009-05

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): ALTU-238
  Interventions: Drug: Somatropin
- 2 (Experimental): ALTU-238
  Interventions: Drug: Somatropin
- 3 (Experimental): ALTU-238
  Interventions: Drug: Somatropin
- 4 (Active Comparator): Nutropin AQ
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — ALTU-238 0.3 mg/kg daily
  Arms: 1
Drug: Somatropin — ALTU-238 0.6 mg/kg daily
  Arms: 2
Drug: Somatropin — ALTU-238 0.9 mg/kg daily
  Arms: 3
Drug: Somatropin — Nutropin AQ 0.043 mg/kg daily
  Arms: 4

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of ALTU-238 in the treatment of children with growth hormone deficiency who have not yet reached puberty who lack the normal ability to make growth hormone themselves. This study will also test if ALTU-238 works as a weekly treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Assent of subject, if applicable, and written informed consent of parent or legal guardian
2. Diagnosis of GHD as defined by a maximum stimulated GH < 7 ng/mL (μg/L) on two stimulation tests (using any two distinct agents from the following list: arginine, L-dopa, clonidine, insulin, or glucagon); if two documented historical tests are not available,test(s) must be performed during Screening period
3. Available results from one or more historical CT or MRI scans of the head obtained at or following the diagnosis of GHD
4. Chronologic age at Screening of 3 to 13 years (inclusive) for boys and 3 to 12 years(inclusive) for girls
5. Bone age at Screening of ≤ 11 years for boys and ≤ 10 years for girls
6. Pre-pubertal at Screening (Tanner stage 1 for both breast/genitalia and pubic hair
7. For subjects with idiopathic GHD, a Screening height SDS ≤ -2.0 (standardized for chronologic age and sex) there is no height SDS requirement if the subject has organic GHD (as defined by a CNS lesion or insult on a historical CT or MRI scan)
8. Pre-treatment annualized height velocity ≤ median (50th percentile) for chronologic age and sex (based on values for delayed maturers provided in Appendix 4), utilizing Screening height and height obtained 52 ± 13 weeks (i.e. 39 to 65 weeks) prior to Screening
9. Screening IGF-1 SDS for chronologic age and sex < -1
10. If on thyroid hormone replacement therapy, the dose must be stable for at least 6 weeks prior to Screening and the free thyroxine level (T4), TSH, and cortisol must be within the normal range at the Screening visit

Exclusion Criteria:

1. History of any prior rhGH, rhIGF-1, or sex steroid treatment
2. History of treatment with any medications that may affect growth
3. Evidence of active intracranial neoplasm per recent serial CT or MRI scans of the head or other criteria
4. Surgery/chemotherapy/radiation therapy for intracranial neoplasm within the prior 52 weeks
5. Any history of non-intracranial neoplasm
6. History of or active benign intracranial hypertension
7. High-dose chronic systemic corticosteroid treatment (oral or injected) within prior 13 weeks
8. Acute or severe illness within prior 26 weeks
9. History of diabetes mellitus, anorexia nervosa, cystic fibrosis, chronic severe kidney or liver disease, chronic infectious disease, inborn errors of metabolism, chromosomal disorders, intrauterine growth retardation, or other childhood disease associated with growth failure
10. History of congenital syndromes associated with abnormal growth, including Turner syndrome, Noonan syndrome, Prader-Willi syndrome, etc.
11. History of severe associated pathology affecting growth, including malnutrition,malabsorption, or bone dysplasia
12. History of autoimmune disease
13. Serum ALT or AST ≥ 1.5X ULN
14. Participation in another clinical trial or treatment with any investigational agent (drug or biologic) within 30 days prior to Baseline if the half-life of the agent is known to be ≤ 6 days or within 6 weeks prior to Baseline if the half-life is > 6 days or not known
15. History of any allergic or abnormal reaction to any of the components of the study drugs
16. Any previous or ongoing clinically significant illness, PE findings, or laboratory abnormality that, in the opinion of the Investigator or the Medical Monitor, could prevent the subject from completing the protocol-specified requirements successfully
17. Poor likelihood, in the Investigator's opinion, that the subject will comply with protocol requirements (e.g., uncooperative attitude, inability to return for follow-up visits, history of medical noncompliance) and/or poor likelihood of completing the study

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Mean change in annualized height velocity from pre-treatment to the first 26 weeks of treatment | 26 Weeks

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Nemours Children's Clinic, Orlando, Florida
  - Baystate Medical Centre, Springfield, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Schneider Children's Hospital, New Hyde Park, New York
  - Children's Hospital Medical Centre, Cincinnati, Ohio
  - Cook Children's Hospital, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington